CLINICAL TRIAL: NCT00163670
Title: The Impact of Sleep Disorders on Motor Vehicle Accidents
Status: Completed | Type: Observational
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: 98/05
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2005-09

CONDITIONS: Sleep Disorders
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Motor vehicle accident
- Control

SUMMARY:
Patients who have sleep disorders may be involved in accidents more frequently than those without. In addition patients who have sleep disorders may have more serious accidents and have increased length of stay.We aim to recruit drivers admitted as a result of a motor vehicle accidents and to ascertain the prevalence of sleep disorders in this group.

ELIGIBILITY:
Inclusion Criteria:Drivers admitted as result of motor vehicle accidents -

Exclusion Criteria:Drivers aged < 18 years

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Naughton, MD,FRACP, Principal Investigator — The Alfred